CLINICAL TRIAL: NCT00288548
Title: Pulmonary Effects of the Combination of Metoprolol and Formoterol in COPD
Brief Title: Metoprolol and Formoterol in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martini Hospital Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MeFCo2
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2006-02-20 (Estimated); Status verified 2006-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Metoprolol

INTERVENTIONS:
Drug: Metoprolol

SUMMARY:
We want to study the effect of the combination of metoprolol (a beta-blocker) with formoterol (a beta-agonist) on long function in patients with Chronic Obstructive Pulmonary Disease (COPD). There are more and more clues that a beta-blocker, when well chosen and in the right dosage, won't harm the long function in patients with COPD. Since a beta-blocker can be a valuable addition to treating patients with heart problems we would like to see if this category of medication can be available for COPD patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* male/female aged between 40-70 inclusive
* COPD defined by GOLD criteria
* FEV1 greater or equal to 60% of predicted without medication
* baseline FEV1 greater or equal than 1.2L
* 10 or more pack years
* no hard contraindications for use of beta blockers
* being able to perform technically acceptable pulmonary function tests
* signed informed consent
* systolic blood pressure equal to 130 or greater

Exclusion Criteria:

* instable COPD during the month before visit 1
* usage of corticosteroids during the month before visit 1
* significant pulmonary diseases other than COPD
* a history of cancer within the last 5 years (basal cell carcinoma or cutaneous squamous cell carcinoma allowed)
* a recent history of myocardial infarction
* use of an investigational drug within one month or six half lives (which ever is greater) of visit 1
* contra-indications for the use of ipratropium-bromide

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2006-02

PRIMARY OUTCOMES:
Difference in airway reactivity after treatment with metoprolol compared to placebo.

SECONDARY OUTCOMES:
Effect of formoterol on airway reactivity comparing metoprolol with placebo.
Borg-scores during provocation test
Peak-flow measurements
CCQ-scores
Exacerbation rate and rescue medication use

CONTACTS AND LOCATIONS:
Overall Officials: René Aalbers, MD, PhD, Principal Investigator — Martini Hospital Groningen
Locations (1):
- Martini Hospital, Groningen, Provincie Groningen, Netherlands